CLINICAL TRIAL: NCT04830072
Title: Mobile Phone Based Personalized and Interactive Augmented Reality (AR) Pictures on Enhancing Brief Advice Model for Smoking Cessation: a Pilot Randomized Controlled Trial
Brief Title: AR Enhanced Pictorial Warnings on Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pictorial warning AR
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; randomized controlled trial; augmented reality; mobile health
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR group (Experimental): Brief AWARD advice + active referral + leaflet + 3 months chat-based support with AR pictures
  Interventions: Behavioral: Brief AWARD advice and active referral to somking cessation services; Behavioral: Chat-based support through Instant Messaging apps; Other: Leaflet; Behavioral: AR images
- Control group (Active Comparator): Brief AWARD advice + active referral + leaflet + 3 months chat-based support
  Interventions: Behavioral: Brief AWARD advice and active referral to somking cessation services; Behavioral: Chat-based support through Instant Messaging apps; Other: Leaflet

INTERVENTIONS:
Behavioral: Brief AWARD advice and active referral to somking cessation services — The AWARD advice includes: (1) Ask about smoking history; (2) Warn about the high risk of smoking; (3) Advise to quit or reduce smoking as soon as possible; (4) Refer smokers to smoking cessation services (with a referral card); (5) Do it again: to repeat the intervention.
Behavioral: Chat-based support through Instant Messaging apps — Participants in the intervention group will receive 3 months of chat-based support through Instant Messaging apps (e.g., WhatsApp, WeChat). The support mainly includes (1) regular messages on health warnings, benefits and methods of quitting, coping craving approach, and promotion to use the SC services; (2) real-time, personalized, and interactive behavioral and psychosocial support through Instant Messaging apps.
Other: Leaflet — Leaflet on harms of smoking
Behavioral: AR images — AR images of the harms of smoking and the benefit of abstinence.
  Arms: AR group

SUMMARY:
This pilot randomized controlled trail aims to test the effects of AR enhanced pictorial effects in harms of smoking and benefit of smoking cessation.

DETAILED DESCRIPTION:
Conventional health warnings on smoking harms mostly include pictures showing smoking consequences such as lung diseases, peripheral vascular diseases, aging, skin lesions, and benefit of quitting such as improved cardiopulmonary functions, skin conditions and risk of diseases, etc. The effects of the information are limited by the generic messages, unattractive images, and lack of interaction. This proposal aims to enhance the "Warn" and "Advice" materials using mobile phone-based augmented reality (AR) technologies to provide personalized, interactive, and attractive images to encourage smokers to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong adults aged 18 or above;
* Smoke at least 1 cigarette daily in the past 30 days;
* Own a smartphone and familiar with instant messaging apps;
* Able to read and communicate in Chinese.

Exclusion Criteria:

* Participate in other smoking cessation services or projects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Self-reported past 7-day point prevalence abstinence | 3 months after baseline
  Abstain from smoking in the past 7 days

SECONDARY OUTCOMES:
Self-reported past 7-day point prevalence abstinence | 1 months after baseline
  Abstain from smoking in the past 7 days
Self-reported smoking reduction by at least 50% | 3 months after baseline
  Defined by at least 50% reduction in baseline daily cigarette consumption
Self-reported smoking reduction by at least 50% | 1 months after baseline
  Defined by at least 50% reduction in baseline daily cigarette consumption
Self-reported quit attempts | 3 months after baseline
  Defined by abstinence for at least 24 hours
Self-reported quit attempts | 1 months after baseline
  Defined by abstinence for at least 24 hours
Recall of pictorial warnings | 3 months after baseline
  Defined by the recall of the quitline on warning pictures
Recall of pictorial warnings | 1 months after baseline
  Defined by the recall of the quitline on warning pictures
Attention of pictorial warnings | 1 months after baseline
  Defined by notice of pictorial warning
Attention of pictorial warnings | 3 months after baseline
  Defined by notice of pictorial warning
Self-reported intention to quit | 1 months after baseline
  Defined by readiness to quit in 30 days
Self-reported intention to quit | 3 months after baseline
  Defined by readiness to quit in 30 days
Reactions to the pictorial warnings | 3 months after baseline
  Defined by behaviors to avoid seeing pictorial warnings
Reactions to the pictorial warnings | 1 months after baseline
  Defined by behaviors to avoid seeing pictorial warnings
Perceived effectiveness of AR images | 1 months after baseline
  Defined by ratings on the effectiveness of AR images to encourage quitting
Perceived effectiveness of AR images | 3 months after baseline
  Defined by ratings on the effectiveness of AR images to encourage quitting

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No